CLINICAL TRIAL: NCT06242197
Title: Comparing the Effectiveness of Written Advice VS. Standard Verbal Advice in Transferring Knowledge to First Degree Relatives of Colorectal Cancer Patients
Brief Title: Comparing the Effectiveness of Written Vs Verbal Advice for First Degree Relatives of Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Thippawan Saengnoi, Doctor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: COA. MURA2023/311
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; First degree relative; Cancer screening; Colonoscopy screening; Family history of colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- written advice (Experimental): written advice (in leaflet form) was given to CRC patients to give to first degree relatives, or send to first degree relatives directly. this leaflet contained information about cancer risk and recommended screening methods.
  Interventions: Other: written advice
- standard verbal advice (Active Comparator): verbal advice about cancer risk and screening methods was given to CRC patients to pass on to their first degree relatives
  Interventions: Other: written advice

INTERVENTIONS:
Other: written advice — written advice (in leaflet form) was given to CRC patients to give to first degree relatives, or send to first degree relatives directly. this leaflet contained information about cancer risk and recommended screening methods.

SUMMARY:
CRC patients were enrolled and asked about their FDR contacts These FDRs were telephoned and enrolled and randomized to receive either written advice and verbal advice about their cancer risk and screening methods. These FDRs were telephoned after 2 weeks to evaluate their knowledge about CRC risk and method of screening to see which method of giving advice was better.

DETAILED DESCRIPTION:
1. Colorectal cancer patients in a tertiary referral hospital who had first degree relatives in the screening range were enrolled into the study.
2. CRC patients and their FDRs were randomized after enrollment into written advice and verbal advice arms
3. CRC patients were asked to give the documents or verbal advice to FDR within 2 wks.
4. A telephone check was done to see if CRC patients had given or sent the advice their FDR.
5. FDR were telephoned to see if they received the document and assessed their knowledge of FDR risk, screening methods, previous screening and other knowledge about CRC.
6. FDRs were given information over the telephone about CRC risk and screening and then asked whether they wanted to have screening or not.

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives of patient with colorectal cancer

Exclusion Criteria:

* First degree relatives whom already diagnosed of colorectal cancer
* First degree relatives whom have colorectal cancer from genetic disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of written advice VS. standard verbal advice in transferring knowledge to first degree relatives of colorectal cancer patients | 3 weeks
  Result of questionnaire about knowing their increase cancer risk

SECONDARY OUTCOMES:
Ascertaining the problem of communicating medical advice between patient and first degree relatives | 3 weeks
  Questionnaire-interview
Determining the knowledge level about colorectal cancer in first degree relatives of CRC patients | 3 weeks
  Questionnaire-interview

CONTACTS AND LOCATIONS:
Overall Officials: Thippawan saengnoi, Ph.D, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramanthibodi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karahalios A, Simpson JA, Baglietto L, MacInnis RJ, Hodge AM, Giles GG, English DR. Change in weight and waist circumference and risk of colorectal cancer: results from the Melbourne Collaborative Cohort Study. BMC Cancer. 2016 Feb 25;16:157. doi: 10.1186/s12885-016-2144-1. PMID 26917541
- [Background] O'Reilly M, Linehan A, Krstic A, Kolch W, Sheahan K, Winter DC, Mc Dermott R. Oncotherapeutic Strategies in Early Onset Colorectal Cancer. Cancers (Basel). 2023 Jan 16;15(2):552. doi: 10.3390/cancers15020552. PMID 36672501
- [Background] Fedirko V, Tramacere I, Bagnardi V, Rota M, Scotti L, Islami F, Negri E, Straif K, Romieu I, La Vecchia C, Boffetta P, Jenab M. Alcohol drinking and colorectal cancer risk: an overall and dose-response meta-analysis of published studies. Ann Oncol. 2011 Sep;22(9):1958-1972. doi: 10.1093/annonc/mdq653. Epub 2011 Feb 9. PMID 21307158
- [Background] Song M, Emilsson L, Roelstraete B, Ludvigsson JF. Risk of colorectal cancer in first degree relatives of patients with colorectal polyps: nationwide case-control study in Sweden. BMJ. 2021 May 4;373:n877. doi: 10.1136/bmj.n877. PMID 33947661
- [Background] Lowery JT, Ahnen DJ, Schroy PC 3rd, Hampel H, Baxter N, Boland CR, Burt RW, Butterly L, Doerr M, Doroshenk M, Feero WG, Henrikson N, Ladabaum U, Lieberman D, McFarland EG, Peterson SK, Raymond M, Samadder NJ, Syngal S, Weber TK, Zauber AG, Smith R. Understanding the contribution of family history to colorectal cancer risk and its clinical implications: A state-of-the-science review. Cancer. 2016 Sep 1;122(17):2633-45. doi: 10.1002/cncr.30080. Epub 2016 Jun 3. PMID 27258162
- [Background] Butterworth AS, Higgins JP, Pharoah P. Relative and absolute risk of colorectal cancer for individuals with a family history: a meta-analysis. Eur J Cancer. 2006 Jan;42(2):216-27. doi: 10.1016/j.ejca.2005.09.023. Epub 2005 Dec 9. PMID 16338133
- [Background] Wilkinson AN, Lieberman D, Leontiadis GI, Tse F, Barkun AN, Abou-Setta A, Marshall JK, Samadder J, Singh H, Telford JJ, Tinmouth J, Leddin D. Colorectal cancer screening for patients with a family history of colorectal cancer or adenomas. Can Fam Physician. 2019 Nov;65(11):784-789. PMID 31722908
- [Background] Tung SY, Wu CS. Risk factors for colorectal adenomas among immediate family members of patients with colorectal cancer in Taiwan: a case-control study. Am J Gastroenterol. 2000 Dec;95(12):3624-8. doi: 10.1111/j.1572-0241.2000.03380.x. PMID 11151903
- [Background] Courtney RJ, Paul CL, Carey ML, Sanson-Fisher RW, Macrae FA, D'Este C, Hill D, Barker D, Simmons J. A population-based cross-sectional study of colorectal cancer screening practices of first-degree relatives of colorectal cancer patients. BMC Cancer. 2013 Jan 10;13:13. doi: 10.1186/1471-2407-13-13. PMID 23305355
- [Background] Fuchs CS, Giovannucci EL, Colditz GA, Hunter DJ, Speizer FE, Willett WC. A prospective study of family history and the risk of colorectal cancer. N Engl J Med. 1994 Dec 22;331(25):1669-74. doi: 10.1056/NEJM199412223312501. PMID 7969357
- [Background] Monahan KJ, Bradshaw N, Dolwani S, Desouza B, Dunlop MG, East JE, Ilyas M, Kaur A, Lalloo F, Latchford A, Rutter MD, Tomlinson I, Thomas HJW, Hill J; Hereditary CRC guidelines eDelphi consensus group. Guidelines for the management of hereditary colorectal cancer from the British Society of Gastroenterology (BSG)/Association of Coloproctology of Great Britain and Ireland (ACPGBI)/United Kingdom Cancer Genetics Group (UKCGG). Gut. 2020 Mar;69(3):411-444. doi: 10.1136/gutjnl-2019-319915. Epub 2019 Nov 28. PMID 31780574
- [Background] Sung JJ, Ng SC, Chan FK, Chiu HM, Kim HS, Matsuda T, Ng SS, Lau JY, Zheng S, Adler S, Reddy N, Yeoh KG, Tsoi KK, Ching JY, Kuipers EJ, Rabeneck L, Young GP, Steele RJ, Lieberman D, Goh KL; Asia Pacific Working Group. An updated Asia Pacific Consensus Recommendations on colorectal cancer screening. Gut. 2015 Jan;64(1):121-32. doi: 10.1136/gutjnl-2013-306503. Epub 2014 Mar 19. PMID 24647008
- [Background] Gimeno-Garcia AZ, Hernandez-Alvarez-de-Buylla N, Nicolas-Perez D, Carrillo M, Hernandez G, Quintero E. Colorectal cancer screening in the familial risk population: Is colonoscopy still the strategy of choice? Gastroenterol Hepatol. 2016 May;39(5):352-60. doi: 10.1016/j.gastrohep.2015.09.009. Epub 2015 Nov 4. PMID 26547615
- [Background] Tsai MH, Xirasagar S, Li YJ, de Groen PC. Colonoscopy screening among US adults aged 40 or older with a family history of colorectal cancer. Prev Chronic Dis. 2015 May 21;12:E80. doi: 10.5888/pcd12.140533. PMID 25996988
- [Background] Hatamian S, Hadavandsiri F, Momenimovahed Z, Salehiniya H. Barriers and facilitators of colorectal cancer screening in Asia. Ecancermedicalscience. 2021 Sep 13;15:1285. doi: 10.3332/ecancer.2021.1285. eCollection 2021. PMID 34824608
- [Background] Tan KK, Lim TZ, Chan DKH, Chew E, Chow WM, Luo N, Wong ML, Koh GC. Getting the first degree relatives to screen for colorectal cancer is harder than it seems-patients' and their first degree relatives' perspectives. Int J Colorectal Dis. 2017 Jul;32(7):1065-1068. doi: 10.1007/s00384-017-2818-4. Epub 2017 Apr 13. PMID 28409270
- [Background] Rawla P, Sunkara T, Barsouk A. Epidemiology of colorectal cancer: incidence, mortality, survival, and risk factors. Prz Gastroenterol. 2019;14(2):89-103. doi: 10.5114/pg.2018.81072. Epub 2019 Jan 6. PMID 31616522
- See also: Prevalence of colorectal cancer in Thailand — http://www.nci.go.th/th/File_download/Nci%20Cancer%20Registry/HOSPITAL-BASED%202014.pdf.
- See also: Clinical guideline for CRC screening — http://dx.doi.org/10.14309/ajg.0000000000001122
- See also: Clinical guideline for CRC screening in Thai — http://www.nci.go.th/th/cpg/Cervical_Cancer3.pdf
- See also: Clinical guideline for CRC screening in first degree relatives — http://dx.doi.org/10.1016/j.jclinepi.2005.07.018